CLINICAL TRIAL: NCT04863209
Title: Effect of Osteopathic Techiniques on Intraocular Pressure: a Randomized Double-blind Clinical Trial
Brief Title: Effect of Osteopathic Techiniques on Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodolfo Amoroso Borges, DO, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RBorges
Record Dates: First submitted 2021-04-20; First posted 2021-04-28 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Intraocular Pressure; Osteopathic Manipulative Treatment
Keywords: intraocular pressure; sphenopalatine ganglion; superior cervical ganglion; aqueous humour

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper cervical manipulation group (Experimental): The patient will be in the supine position. The cephalic hand will make contact with one side of the patient's skull, leaving the sternocleidomastoid muscle between the third and fourth fingers. The caudal hand will make global contact with the patient's skull on the opposite side. The therapist should place his torso on the patient's head, leaving the two forearms aligned with the axis of the patient's spine, as this technique is applied to the axis of the odontoid process of the ax. With neutral flexion-extension the therapist will place the rotation parameter to the opposite side (70-80 degrees) and a small contralateral inclination. Then it will search for the driving barrier with a small axial traction movement. When the driving barrier is found, the thrust should be applied in a helical direction, increasing rotation and traction. It will be applied bilaterally.
  Interventions: Other: Upper cervical manipulation
- Sphenopalatine ganglion group (Experimental): The patient will be supine on the bench and the therapist with gloves will sit next to the patient contralateral to the manipulated sphenopalatine ganglion (SPG). One of the therapist's hands will be placed flat in contact with the apex of the patient's head to stabilize it. The patient will be instructed to open his mouth and deviate the mandible laterally to the same side of the ganglion to be treated. The therapist will then apply pressure to the SPG with the fifth finger of your other hand in the patient's mouth, moving up along the alveolar process of the maxilla teeth to reach the pterygoid process. The therapist will keep the patient's head elevated until the lateral pterygoid muscle relaxes. Then, the pressure will be applied into the pterygopalatine fossa. The therapist will then apply gentle pressure on the SPG with the pulp of the fifth finger until tissue relaxation. He will then release the contralateral SPG in the same way.
  Interventions: Other: Sphenopalatine ganglion manipulation
- Control Group (No Intervention): The patient will lie down on the bench for 10 minutes.

INTERVENTIONS:
Other: Upper cervical manipulation — The patient will receive an upper cervical manipulation as described in the Experimental Group 1.
  Arms: Upper cervical manipulation group
Other: Sphenopalatine ganglion manipulation — The patient will receive a sphenopalatine ganglion as described in the Experimental Group 2.
  Arms: Sphenopalatine ganglion group

SUMMARY:
The purpose of this study is to assess the effects osteopathic techniques at the upper cervical vertebrae or at the sphenopalatine ganglia on the intraocular pressure.

DETAILED DESCRIPTION:
The 7 volunteers will be randomized into 3 groups and there will be an experimental group 1 that will receive a technique of manipulation of the upper cervical, an experimental group 2 that will receive a technique of manipulation of the sphenopalatine ganglion and a control group that will not receive any intervention. Each volunteer will participate in the 3 groups. There will be 4 assessments, one before the procedure and one just after each procedure, including the control.

ELIGIBILITY:
Inclusion Criteria:

* Intraocular pressure below 21mmHg

Exclusion Criteria:

* Positive Klein test
* Use of medications that affect the circulatory system in up to one month before the procedures;
* Caffeine use 24 hours before procedures;
* Presence of ophthalmic diseases;
* History of hypertension or diabetes;
* Blindness;
* Tumor in the head;
* Skull or cervical fractures that occurred less than 6 months ago.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Change of the intraocular pressure after upper cervical manipulation | Immediately after the intervention and 30 minutes after the intervention
  After this manipulation, it is expected that there will be a sympathetic response increasing the intraocular pressure.
Change of the intraocular pressure after sphenopalatine ganglion manipulation | Immediately after the intervention and 30 minutes after the intervention
  After this manipulation, it is expected that there will be a parasympathetic response decreasing the intraocular pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Educação Física, Jundiaí, São Paulo, Brazil